CLINICAL TRIAL: NCT05132725
Title: Studying the Effect of Gluten Free Diet Alone Versus Combination of Gluten Free Diet With Either Carbohydrate Count or Dietary Approach to Reduce Hypertension Diet on Their Glycemic Control, Growth Rate and Quality of Life Among Children With Type 1 Diabetes Mellitus and Celiac Disease
Brief Title: Carbohydrate Counting and DASH Intervention Among Children With Diabetes and Celiac Disease.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Jordan (Other)
Responsible Party: Principal Investigator, Marah Al Majali, student, University of Jordan
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UJordanM
Record Dates: First submitted 2021-11-13; First posted 2021-11-24 (Actual); Last update posted 2021-11-24 (Actual); Status verified 2021-11

CONDITIONS: Diabetes Mellitus, Type 1; Celiac Disease in Children
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Diet Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Dietary intervention CHO counting combined with GFD (Experimental): Carbohydrate counting diet will be prepared according to Kulkarni, (2005). Tailored diet plans according to patient's food preference, physical activity level and appropriate insulin: Carbohydrates ratio will be prescribed for each participants. Diets were based on each participants' recommended intakes of energy, protein (15-25%), fat (30-40%) and carbohydrate (40-50%) (Thomas and Gutierrez, 2005; Kleinwechter et al., 2014). Energy requirement will be determined in the participants' weight. The carbohydrate counts will be distributed into three main meals and 3 snacks, with the general dietary advice and diet that will be prescribed by hospital for participants
  Interventions: Behavioral: diet therapy
- Dietary intervention CHO Counting with GFD & DASH (Experimental): The recommended intakes of energy, protein (15-25%), fat (30-40%) and carbohydrate (40-50%) will be similar to that in carbohydrate counting diet which mentioned above. DASH diet food choices will be inserted in the diet of the participants assigned for the combined diet of DASH and carbohydrate counting. The emphasis will be more on the fruits and vegetables group (>8 servings/day), whole grains (at least half of the amount of the total servings of cereals; 6-8 servings/day), fat free dairy products (2-3 servings/day), lean meat and plant proteins (0-2 servings/day) and nuts (5-7 servings/week). From the fat group olive oil will represent the main type of fat (20-25% of total fat %). Adequate intake of sodium (2000mg) will be applied into participants' diet, with the general dietary advice and diet that will be prescribed by hospital for participants
  Interventions: Behavioral: diet therapy
- General Dietary guidlines (No Intervention): the general dietary advice and diet that will be prescribed by hospital for participants

INTERVENTIONS:
Behavioral: diet therapy — Adjusting the quantity and quality of food intake to improve glycemic control, growth rate and quality of life among children with type 1 diabetes and celiac disease.
  Arms: Dietary intervention CHO Counting with GFD & DASH; Dietary intervention CHO counting combined with GFD

SUMMARY:
Study is an interventional clinical trial. children (aged 6-18 years) diagnosed with type 1 diabetes and celiac disease will be recruited conveniently from Endocrinology pediatric clinic at Prince Hamzah Hospital. Amman, Jordan. A sample of 45 diagnosed children, who will meet the inclusion criteria and will be agreed to participate will be centrally randomized to follow carbohydrate counting with GFD dietary intervention, carbohydrate counting with GFD and DASH dietary intervention, and control dietary intervention.

DETAILED DESCRIPTION:
the main objective of this study to compare the effects of three diets: carbohydrate count with gluten-free diet, DASH and carbohydrate count with gluten-free diet, and gluten-free diet alone on glycemic control, growth rate, and the quality of life of 45 individual patients diagnosed with diabetes and celiac disease, who are receiving care in Prince Hamzah Hospital, and aged between 6-18 years, will be enrolled in this study. the duration of the follow-up will be up to ( 9 months); starting from the first interview and enrollment till reaching 9 months from the intervention. all the biochemical tests that are routinely measured will be recorded for each patients during the follow-up duration. these biochemical tests will be, mainly hemoglobin A1C, serum glucose, tissue-trans glutamines IgA( TTG IgA), vitamin D, calcium, phosphorus, and acute intermittent porphyria ( AIP) and will be recorded at baseline, after 6 months and at the end of the study (12 months). growth rate, and quality of life will be also assessed at based line, after 6 months and at the end of the study.

ELIGIBILITY:
Inclusion Criteria: 1- Jordanian children aged between 6 to 18 years old . 2- diagnosed with diabetes type 1 and celiac disease together. -

Exclusion Criteria: 1- any children diagnosed with celiac disease alone. 2- any children diagnosed with type 1 diabetes alone. 3- any children with different disease.

-

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 45 (Estimated)
Dates: Start 2021-11-15 (Estimated); Primary Completion 2022-06-15 (Estimated); Study Completion 2022-11-11 (Estimated)

PRIMARY OUTCOMES:
HbA1c | one year
  Hemoglobin A1c% at both baseline and endline of intervention
glucose serum | one year
  fasting blood glucose% at both baseline and endline of intervention.
TTG-IgA | one year
  TTG-IgA% \ at both and endline of intervention.

SECONDARY OUTCOMES:
Weekly weight gain | one year
  weight in kilogram will be measured every 3 months for all participants.
height | one year
  height will be measured every 3 months for participants.
BMI | one year
  body mass index will be measured according to the weight and height.

CONTACTS AND LOCATIONS:
Overall Officials: marah AT al-majali, master, Principal Investigator — student; reema tayyem, phd, Study Director — supervisor
Locations (1):
- Marah Al Majali, Amman, Jordan

REFERENCES:
- [Background] Agostoni C, Decsi T, Fewtrell M, Goulet O, Kolacek S, Koletzko B, Michaelsen KF, Moreno L, Puntis J, Rigo J, Shamir R, Szajewska H, Turck D, van Goudoever J; ESPGHAN Committee on Nutrition:. Complementary feeding: a commentary by the ESPGHAN Committee on Nutrition. J Pediatr Gastroenterol Nutr. 2008 Jan;46(1):99-110. doi: 10.1097/01.mpg.0000304464.60788.bd. PMID 18162844
- [Background] Ajlouni K, Khader YS, Batieha A, Ajlouni H, El-Khateeb M. An increase in prevalence of diabetes mellitus in Jordan over 10 years. J Diabetes Complications. 2008 Sep-Oct;22(5):317-24. doi: 10.1016/j.jdiacomp.2007.01.004. Epub 2008 Apr 16. PMID 18413210
- [Background] Akobeng AK, Ramanan AV, Buchan I, Heller RF. Effect of breast feeding on risk of coeliac disease: a systematic review and meta-analysis of observational studies. Arch Dis Child. 2006 Jan;91(1):39-43. doi: 10.1136/adc.2005.082016. Epub 2005 Nov 15. PMID 16287899
- [Background] Bjorck S, Brundin C, Karlsson M, Agardh D. Reduced Bone Mineral Density in Children With Screening-detected Celiac Disease. J Pediatr Gastroenterol Nutr. 2017 Nov;65(5):526-532. doi: 10.1097/MPG.0000000000001568. PMID 28319607
- [Background] Caio G, De Giorgio R, Volta U. Coeliac disease and dermatitis herpetiformis. Lancet. 2018 Sep 15;392(10151):916-917. doi: 10.1016/S0140-6736(18)31486-7. No abstract available. PMID 30238885
- [Background] Chander AM, Nair RG, Kaur G, Kochhar R, Dhawan DK, Bhadada SK, Mayilraj S. Genome Insight and Comparative Pathogenomic Analysis of Nesterenkonia jeotgali Strain CD08_7 Isolated from Duodenal Mucosa of Celiac Disease Patient. Front Microbiol. 2017 Feb 2;8:129. doi: 10.3389/fmicb.2017.00129. eCollection 2017. PMID 28210247
- [Background] Dydensborg Sander S, Hansen AV, Stordal K, Andersen AN, Murray JA, Husby S. Mode of delivery is not associated with celiac disease. Clin Epidemiol. 2018 Mar 19;10:323-332. doi: 10.2147/CLEP.S152168. eCollection 2018. PMID 29593435
- [Background] Kaur N, Bhadada SK, Minz RW, Dayal D, Kochhar R. Interplay between Type 1 Diabetes Mellitus and Celiac Disease: Implications in Treatment. Dig Dis. 2018;36(6):399-408. doi: 10.1159/000488670. Epub 2018 Jul 25. PMID 30045024